CLINICAL TRIAL: NCT05127200
Title: Effect of the Neuromodulation of the Cervical Spinal Cord on Nociceptive Processing in Healthy Volunteers - a Randomized, Double-blinded Study
Brief Title: Cervical Neuromodulation and Nociceptive Processing
Acronym: MICROVOLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021/02SEP/359
Record Dates: First submitted 2021-10-05; First posted 2021-11-19 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Nociceptive Pain
Keywords: tsDCS; non-invasive neuromodulation; healthy volunteers
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tsDCS (cervical active, lumbar sham) (Experimental): Participants will receive:
  1. 20 minutes of 2.5 milliampere (mA) anodal tsDCS at the cervical level.
  2. sham tsDCS at the lumbar level.
  Interventions: Device: Starstim (Neuroelectrics)
- Anodal tsDCS (cervical sham, lumbar active) (Active Comparator): Participants will receive:
  1. 20 minutes of 2.5 milliampere (mA) anodal tsDCS at the lumbar level.
  2. sham tsDCS at the cervical level.
  Interventions: Device: Starstim (Neuroelectrics)

INTERVENTIONS:
Device: Starstim (Neuroelectrics) — Anodal transcutaneous spinal direct current stimulation (a-tsDCS)

SUMMARY:
Several studies have demonstrated that direct currents delivered through the skin at the level of the lumbar spinal cord can influence spinal cord function. In human volunteers, anodal lumbar transcutaneous spinal direct current stimulation (tsDCS) alters spinal processing of nociceptive inputs. Whether cervical tsDCS is able to do the same is less well known.

DETAILED DESCRIPTION:
The investigators will compare the effects on the nociceptive processing of healthy volunteers of cervical and lumbar tsDCS. This study will be a double-blinded, sham-controlled, cross-over trial. Each participant will undergo two experimental sessions (anodal cervical tsDCS and sham lumbar tsDCS vs. sham cervical tsDCS and anodal lumbar tsDCS), separated by at least one week.

ELIGIBILITY:
Inclusion Criteria:

- Healthy young adults

Exclusion Criteria:

* Known medical conditions (e.g., diabetes, neuropathy, psychiatric disorders, seizure, migraine, pacemaker or other implanted medical devices...)
* Use of any medication (except contraception)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Change in contact-heat evoked potentials amplitude | Change from Baseline, at 15-minutes after the end of stimulation
  N2/P2 amplitude

SECONDARY OUTCOMES:
Change in intensity of perception to contact-heat nociceptive stimuli | Change from Baseline, at 15-minutes after the end of stimulation
  Difference in temperature (°C) needed to elicit a pain sensation of similar intensity in the upper and lower limb
Change in temporal summation of pain | Change from Baseline, at 15-minutes after the end of stimulation
  Wind-up ratio (WUR) to mechanical pinprick stimuli
Change in intensity of perception to mechanical pinprick nociceptive stimuli | Change from Baseline, at 15-minutes after the end of stimulation
  Numerical rating scale (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: André Mouraux, MD, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- NOCIONS lab, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lenoir C, Jankovski A, Mouraux A. Anodal Transcutaneous Spinal Direct Current Stimulation (tsDCS) Selectively Inhibits the Synaptic Efficacy of Nociceptive Transmission at Spinal Cord Level. Neuroscience. 2018 Nov 21;393:150-163. doi: 10.1016/j.neuroscience.2018.10.007. Epub 2018 Oct 12. PMID 30321585